CLINICAL TRIAL: NCT02391220
Title: The Effect of a Symbiotic LCA Yoghurt on Health-related Quality of Life and the Symptoms of Irritable Bowel Syndrome in Adults: A Randomized, Double-blind, Placebo Controlled, Multicentre Clinical Trial
Brief Title: Assessment of the Symbiotic Fermented Milk in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinres Farmacija d.o.o. (Industry)
Collaborators: Competence Centre for Biotechnology Research and Innovation (Unknown); European Regional Development Fund (Other); Ministry of Education, Science and Sport of the Republic of Slovenia (Unknown); Institute of Dairy Science and probiotics, Biotechnical Faculty, UL (Unknown); Dairy Celeia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KC_BRIN
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symbiotic (Active Comparator): LCA symbiotic fermented milk, 180 g pot, twice daily.
  Interventions: Other: LCA symbiotic fermented milk
- Placebo (Placebo Comparator): heat-treated fermented milk, 180 g pot, twice daily.
  Interventions: Other: heat-treated fermented milk

INTERVENTIONS:
Other: LCA symbiotic fermented milk — LCA symbiotic fermented milk with the probiotic cultures Lactobacillus acidophilus La-5® and Bifidobacterium animalis ssp. lactis BB-12® and the Beneo dietary fibers.
  Arms: Symbiotic
Other: heat-treated fermented milk — heat-treated fermented milk without probiotic cultures and dietary fibres
  Arms: Placebo

SUMMARY:
This study evaluates the effect of a symbiotic fermented milk on health-related quality of life and irritable bowel syndrome (IBS) symptoms in patients with constipation-predominant IBS.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is one of the most common digestive disorders in the developed world which. It is associated to numerous symptoms, of which the most characteristic are recurrent pain or discomfort in the abdominal region, changes and difficulties related to bowel movements, and bloating. Although not dangerous, the disease may significantly impair the patients' quality of life. Treatment is symptomatic, but currently not very efficient. The use of probiotics in the treatment of IBS is a promising approach and has been the subject of much research in the last two decades.

The purpose of this randomized, placebo-controlled study is to assess changes in health-related quality of life in patients with constipation-predominant IBS after regular consumption of symbiotic fermented milk (containing probiotics and dietary fibres) and to assess its effects on some symptoms, like abdominal pain or discomfort, bloating, and chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed constipation-predominant irritable bowel syndrome (on the basis of Rome III criteria) (≥ 25 % lumpy or hard stools and ≤ 25 % mushy or watery stools).
* Meeting Rome III criteria for the determination of irritable bowel syndrome in the last 6 months prior to inclusion and the presence of symptoms such as abdominal pain, bloating and general digestive discomfort at least twice a week in the last 3 months prior to inclusion.
* Colonoscopy in the last 7 years prior to inclusion with normal results.

Exclusion Criteria:

* Diarrhoea-predominant irritable bowel syndrome (≥ 25 % mushy or watery stools and ≤ 25 % lumpy or hard stools).
* Clinical signs of alarm, such as rectorrhagia, fever, recent unexplained weight loss.
* Organic gastrointestinal diseases, including chronic inflammatory bowel disease and systemic diseases with gastrointestinal difficulties.
* Severe abdominal pain and the taking of analgesics or antispasmodics for the previous 5 days or more.
* Having begun treatment with psychotropic medicines or other drugs for the treatment of irritable bowel syndrome within the previous month.
* Dietary habits that could influence the assessment of the investigational product, such as slimming or a vegetarian diet.
* Known allergy to ingredient(s) in the investigational product.
* Known medical or psycho-physical condition that is, in the opinion of the investigator, in conflict with consumption of the investigational product and/or the course of the study.
* Participation in another clinical study less than one month before inclusion or concurrent participation in another clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Quality of life | 4 weeks of product consumption
  assessed by IBS-QoL questionnaire

SECONDARY OUTCOMES:
Improvements in IBS symptoms (bloating, abdominal pain, satisfaction with bowel movement, stool frequency and stool consistency) | 4 weeks of product consumption
  assessed by IBS - Severity Scoring System
Improvements in IBS symptoms (bloating, abdominal pain, satisfaction with bowel movement, stool frequency and stool consistency) | 2 weeks of product consumption
  assessed by IBS - Severity Scoring System
Quality of life | 2 weeks of product consumption
  assessed by IBS-QoL questionnaire